CLINICAL TRIAL: NCT07328711
Title: Study on Novel Immunomodulatory Therapeutic Regimens for Clinical Cure of Chronic Hepatitis B and Efficacy Prediction
Brief Title: Immunomodulatory Therapy and Predictors of Clinical Cure in Chronic Hepatitis B
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Bo Feng, Dr., Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202424084
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-05

CONDITIONS: Chronic Hepaititis B
Keywords: hepatitis B immunoglobulin; functional cure
MeSH Terms: interventions — hepatitis B hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBIG immunization group (Experimental): Patients with HBsAg seroclearance will receive an intramuscular injection of HBIG 400 IU upon enrollment. Based on the results of the hepatitis B serology panel follow-up, a supplemental HBIG injection will be administered promptly when necessary (i.e., when anti-HBs is negative or anti-HBs < 100 mIU/mL), with the goal of achieving anti-HBs seroconversion and maintaining its level above 100 mIU/mL.
  Interventions: Drug: Hepatitis B Immunoglobulin (HBIg)
- control group (No Intervention)

INTERVENTIONS:
Drug: Hepatitis B Immunoglobulin (HBIg) — Patients with HBsAg seroclearance will receive an intramuscular injection of HBIG 400 IU upon enrollment. Based on the results of the hepatitis B serology panel follow-up, a supplemental HBIG injection will be administered promptly when necessary (i.e., when anti-HBs is negative or anti-HBs < 100 mIU/mL), with the goal of achieving anti-HBs seroconversion and maintaining its level above 100 mIU/mL.
  Arms: HBIG immunization group

SUMMARY:
Achieving clinical cure, defined as hepatitis B surface antigen (HBsAg) seroclearance, represents a major research focus and an ideal therapeutic goal for chronic hepatitis B (CHB). A significant challenge in CHB management lies in promoting clinical cure, reducing relapse, and progressing towards complete cure. Studies have found that in patients who achieve HBsAg seroclearance following peginterferon alfa (PegIFNα) therapy, the seroconversion of anti-HBs and its attainment to a certain level are crucial for minimizing relapse. Strategies to promote anti-HBs seroconversion include active immunization (hepatitis B vaccine) and passive immunization (hepatitis B immunoglobulin, HBIG). Existing literature and preliminary findings from our team suggest that hepatitis B vaccine alone is ineffective in preventing relapse after clinical cure. This project proposes a multicenter, prospective, randomized controlled study. It will enroll CHB patients who have achieved HBsAg seroclearance with PegIFNα-based therapy, with the primary endpoint being the sustained HBsAg seroclearance rate at 48 weeks. The study will compare the efficacy between a group receiving HBIG immunization and a non-immunization control group. We anticipate that passive immunization with HBIG following HBsAg seroclearance will lead to a sustained clinical cure in CHB patients. This study aims to explore novel approaches for reducing relapse after clinical cure and pursuing complete cure, identify relevant biomarkers, and establish corresponding predictive models.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 60 years (inclusive).
2. Documented HBsAg and/or HBV DNA positivity for over 6 months.
3. Achieved HBsAg seroclearance (<0.05 IU/mL) following a PegIFNα-based treatment regimen.
4. HBeAg negative and HBV DNA <10 IU/mL.
5. Good compliance and willingness to voluntarily sign the informed consent form.

Exclusion Criteria:

1. Current decompensated cirrhosis or a history of decompensated cirrhosis.
2. Individuals with spontaneous or Nucleos(t)ide analogue-induced HBsAg seroclearance.
3. Coinfection with other viruses, such as hepatitis A, C, D, E viruses, or human immunodeficiency virus (HIV).
4. Severe concurrent physical or mental illnesses other than hepatitis B, including uncontrolled primary renal, cardiac, pulmonary, vascular, neurological, digestive, or severe metabolic diseases (e.g., uncontrolled hyperthyroidism, severe diabetic complications, adrenal disorders), immunodeficiency diseases, or severe infections; active or suspected malignancy, or a history of malignancy.
5. Use of corticosteroids, immunosuppressants, or chemotherapeutic agents within the 6 months prior to enrollment or at present.
6. Concurrent other liver diseases such as alcoholic liver disease or autoimmune liver disease.
7. Body Mass Index (BMI) > 28 kg/m².
8. Any other condition considered by the investigator to potentially compromise patient compliance or otherwise make the patient unsuitable for participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The sustained HBsAg seroclearance rate (HBsAg < 0.05 IU/mL) at 48 weeks after initial HBsAg seroclearance | From enrollment to 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided